CLINICAL TRIAL: NCT00816972
Title: Pilot Efficacy and Safety Field Trial of Desloratadine Administered Concomitantly With Oxybutynin, in Subjects With Seasonal Allergic Rhinitis and Post-Nasal Drip
Brief Title: Desloratadine With Oxybutynin for the Treatment of Seasonal Allergic Rhinitis and Post-Nasal Drip (Study P04258)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04258
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Post-nasal Drip; Seasonal Allergic Rhinitis; Rhinorrhea
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinorrhea | interventions — desloratadine; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- DL 2.5 mg (Active Comparator): Desloratadine 2.5 mg twice daily (BID) + Placebo for Oxybutynin 2.5 mg BID for 7 days
  Interventions: Drug: Desloratadine 2.5 mg; Drug: Placebo for Oxybutynin 2.5 mg
- OXY 5 mg (Active Comparator): Placebo for Desloratadine 2.5 mg BID + Oxybutynin 5 mg BID for 7 days
  Interventions: Drug: Oxybutynin 2.5 mg; Drug: Placebo for Desloratadine 2.5 mg
- DL 2.5 mg + OXY 2.5 mg (Experimental): Desloratadine 2.5 mg BID + Oxybutynin 2.5 mg BID + Placebo for Oxybutynin 2.5 mg BID for 7 days
  Interventions: Drug: Desloratadine 2.5 mg; Drug: Oxybutynin 2.5 mg; Drug: Placebo for Oxybutynin 2.5 mg
- DL 2.5 mg + OXY 5 mg (Experimental): Desloratadine 2.5 mg BID + Oxybutynin 5 mg BID for 7 days
  Interventions: Drug: Desloratadine 2.5 mg; Drug: Oxybutynin 2.5 mg
- Placebo (Placebo Comparator): Placebo for Desloratadine 2.5 mg BID + Placebo for Oxybutynin 2.5 mg BID for 7 days
  Interventions: Drug: Placebo for Desloratadine 2.5 mg; Drug: Placebo for Oxybutynin 2.5 mg

INTERVENTIONS:
Drug: Desloratadine 2.5 mg — Desloratadine 2.5 mg BID
  Other Names: SCH 034117; Clarinex
  Arms: DL 2.5 mg; DL 2.5 mg + OXY 2.5 mg; DL 2.5 mg + OXY 5 mg
Drug: Oxybutynin 2.5 mg — Oxybutynin 2.5 mg BID
  Other Names: Ditropan
  Arms: DL 2.5 mg + OXY 2.5 mg; DL 2.5 mg + OXY 5 mg; OXY 5 mg
Drug: Placebo for Desloratadine 2.5 mg — Placebo BID
  Arms: OXY 5 mg; Placebo
Drug: Placebo for Oxybutynin 2.5 mg — Placebo BID
  Arms: DL 2.5 mg; DL 2.5 mg + OXY 2.5 mg; Placebo

SUMMARY:
This was a 1-week study of desloratadine (DL) plus oxybutynin (OXY) at two dose levels in the treatment of post-nasal drip in participants with seasonal allergic rhinitis. Participants received either desloratadine twice a day, oxybutynin twice a day, desloratadine plus lower-dose oxybutynin twice a day, desloratadine plus higher-dose oxybutynin twice a day, or placebo for 7 days.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* be >=18 years of age,
* be free of any clinically significant disease that would interfere with study, other than seasonal allergic rhinitis (SAR),
* have a documented diagnosis of SAR for >=2 years,
* have had a positive skin-prick test,
* be sufficiently symptomatic at the Screening visit,
* for the 3 calendar days immediately prior to baseline visit, plus the AM of the baseline visit, the seven twice-daily run-in diary PRIOR total nasal symptom scores must have totaled >=42, the Total Non-Nasal Symptoms score must have totaled >=28, and the total Post Nasal Drip score must have totaled >=14,
* be in general good health.

Exclusion Criteria:

Subjects who have:

* certain medical conditions or medical histories,
* allergies to any of the components in any of the study medications,
* nasal structure abnormalities,
* dependency to nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids,
* used any investigational drug use in past 30 days,
* received immunotherapy (desensitization)
* are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2005-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean daily AM/PM Prior post-nasal drip scores averaged over the entire treatment period | Days 1 to 7 +/- 2 days

SECONDARY OUTCOMES:
Anterior rhinorrhea averaged over Days 1 to 8 | Days 1 to 8